CLINICAL TRIAL: NCT05768308
Title: Effectiveness and Mediators of Change of an Online CBT Intervention for Students With Adjustment Disorder - Study Protocol for a Randomized Controlled Trial
Brief Title: Online CBT Intervention for Students With Adjustment Disorder
Acronym: Online CBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Juszczyk, Msc Aleksandra Juszczyk-Kalina, University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/01/2023
Record Dates: First submitted 2023-02-13; First posted 2023-03-14 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Adjustment Disorders
Keywords: adjustment disorder; students; internet psychological interventions; cognitive behavioural therapy
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet CBT-UP intervention (iCBT-UP) (Experimental): Patricipants in the experimental group will receive online cbt intervention for students with adjustment disorder (iCBT-UP).
  Interventions: Behavioral: Internet CBT-UP intervention iCBT-UP
- Internet Progressive Muscle Realxation Training (iPMR) (Active Comparator): Participants from the active control group will receive progressive muscle relaxation training (iPMR).
  Interventions: Behavioral: Internet Progressive Muscle Realxation Training (iPMR)
- Waiting List (No Intervention): Participants from the waiting list condition will receive access to the choosen intervention after 6-weeks waiting period.

INTERVENTIONS:
Behavioral: Internet CBT-UP intervention iCBT-UP — The self-helped internet intervention for students experiencing emotional difficulties, especially adjustment disorder. This intervention is based on transdiagnostic cbt principles - unified protocol (Barlow et al., 2018). It is a modular intervention consisting of six modules teaching different skills of dealing with emotions. Intervention is interactive and contains of video materials, quizes, texts and audio materials.
  Arms: Internet CBT-UP intervention (iCBT-UP)
Behavioral: Internet Progressive Muscle Realxation Training (iPMR) — Participants from the active control group will receive progressive muscle relaxation training (iPMR) (Bernstein, Borkovec, Hazlett-Stevens, 2000). It is also a modular intervention and, similar to the i-cbt condition, consists of 5 modules. During the intervention, participants learn how to progressively tighten and relax different muscle groups.The first module is planned for two weeks and the rest of them for one week each. Intervention consists of video materials and audio guided relaxations. Participants are encouraged to train these relaxations once a day.
  Arms: Internet Progressive Muscle Realxation Training (iPMR)

SUMMARY:
The aim of this study is to evaluate the effectiveness of online cognitive-behavioral intervention based on Unified Protocol and mediators of obtained changes among polish students with adjustment disorder. The intervention is fully self-helped and based on Unified Protocol principles. Control conditions contain of online progressive muscle relaxation group and waiting list.

DETAILED DESCRIPTION:
Adjustment problems are highly prevalent among students around the world (Conley et.al., 2013). Unfortunately only half of students in need receive psychological help (Eisenberg et al., 2018). For these reasons, there is a need to develop and evaluate new, more scalable forms of treatment for students with adjustment disorder - such as internet therapeutic programs. Therefore the aim of the present research is to evaluate the effectiveness of online cognitive-behavioural therapy intervention. Mediators of obtained changes will also be evaluated. The present study has a potential for the development of a scalable, well researched treatment option for students experiencing adjustment disorder - internet psychological intervention.

ELIGIBILITY:
Inclusion Criteria:

* having a student status
* 18 years old or older,
* having access to the internet and using computer or smartphone,
* meeting the diagnostic criteria of adjustment disorder based on a total sum score > 47,5 in ADNM-20 questionnaire
* meeting diagnostic criteria for AjD in MINI Interview.

Exclusion Criteria:

* an increased risk of suicidality intent or ideation (at least moderate scores on the MINI and/or a score > 2 on item 9 from the PHQ-9),
* psychotic disorder, eating disorder, anti-social personality disorder and/or alcohol/substance use disorder as indicated by the MINI
* receiving another psychological treatment at the start of the study
* having no time for participation in program
* receiving pharmacological psychiatric treatment not stabilized 6 weeks prior the start of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in Adjustment disorder | measured at baseline, immediately after the interventions and 1 month follow up
  Adjustment disorder - The Adjustment Disorder New Module 20 (ADNM-20)

SECONDARY OUTCOMES:
Change in Depression | measured at baseline, immediately after the interventions and 1 month follow up
  The patient health questionnaire-9 (PHQ-9)
Change in General Anxiety Disorder | measured at baseline, immediately after the interventions and 1 month follow up
  General Anxiety Disorder-7 (GAD-7)
Change in Stress | measured at baseline, immediately after the interventions and 1 month follow up
  Scale of experienced stress (PSS-10)
Change in Satisfaction with life | measured at baseline, immediately after the interventions and 1 month follow up
  Satisfaction with life scale (SWLS)
Change in Academic Adjustment | measured at baseline, immediately after the interventions and 1 month follow up
  Academic adjustment scale (AAS)
Change in Experiential Avoidance | measured at baseline, immediately after the interventions and 1 month follow up
  Acceptance and Action Questionnaire
Change in Cognitive Fusion | measured at baseline, immediately after the interventions and 1 month follow up
  Cognitive Fusion Questionnaire (CFQ)
Change in Self-compassion | measured at baseline, immediately after the interventions and 1 month follow up
  Self Compassion Scale - Short Form (SCS-SF)
Change in Mindfulness | measured at baseline, immediately after the interventions and 1 month follow up
  Five Facet Mindfulness Questionnaire (FFMQ-15)
Change in Persevative thinking | measured at baseline, immediately after the interventions and 1 month follow up
  Perseverative Thinking Questionnaire (PTQ)
Change in Mental well-being | measured at baseline, immediately after the interventions and 1 month follow up
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
Change in Cognitive functioning | measured at baseline, immediately after the interventions and 1 month follow up
  Stroop Task (color-word)
Change in Academic performance | measured at baseline, immediately after the interventions and 1 month follow up
  This index will be based on a three recently received grades. The mean will be assessed.
Change in Daily Depressogenic adjustment | 7 days during the first week of the intervention and 7 days during the sixth week of the intervention time
  Measured in daily diaries. It will be measured by three items based on Becks triad.
Change in Daily negative thinking | 7 days during the first week of the intervention and 7 days during the sixth week of the intervention time
  Measured in daily diaries. Rumination and worrying. Daily worry measures will be measured with three items taken from Meyer et al. (1990).
Change in Emotional regulation | 7 days during the first week of the intervention and 7 days during the sixth week of the intervention time
  Measured in daily diaries. cognitive restructuring and emotional supression. This variables will be measured using one item (each scale) from Emotional Regulation Questionnaire (ERQ).
Change in Self-compassion | 7 days during the first week of the intervention and 7 days during the sixth week of the intervention time
  Measured in daily diaries, by three items from Self Compassion Scale (SCS).
Change in Daily-affect | 7 days during the first week of the intervention and 7 days during the sixth week of the intervention time
  Measured in daily diaries, based on circumplex model.
Change in Procrastination | 7 days during the first week of the intervention and 7 days during the sixth week of the intervention time
  Measured in daily diaries, by three items from The Pure Procrastination scale.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Juszczyk-Kalina, Msc, Principal Investigator — University of Warsaw

REFERENCES:
- [Derived] Juszczyk-Kalina A, Holas P, Farchione TJ. Effectiveness and mediators of change of an online CBT intervention for students with adjustment disorder-study protocol for a randomized controlled trial. Trials. 2023 Dec 1;24(1):777. doi: 10.1186/s13063-023-07744-9. PMID 38041148